CLINICAL TRIAL: NCT03501420
Title: Patient Phenotypes and Treatment Pathways in Primary Sjogren's Syndrome: an International Cross-sectional Survey of Rheumatologists and Adult Primary Sjögren's Syndrome Patients With Systemic Involvement (Adelphi 2018 pSS Disease Specific Programme)
Brief Title: Adelphi Primary Sjogren's Syndrome (pSS) Disease Specific Programme (DSP)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Adelphi Real World (Industry)
Responsible Party: Sponsor
Other Study IDs: 207382
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Sjogren's Syndrome
Keywords: Belimumab; Disease Specific Programme; rheumatologist; Benlysta; Primary Sjögren's Syndrome; Adelphi pSS DSP
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians: A sample of 230 to 325 rheumatologists actively involved in management and treatment decisions of pSS subjects in France, Italy, Spain, Germany and the United States will be included in the survey.
  Interventions: Other: Interview; Other: PRFs
- Subjects with pSS: Subjects with a confirmed diagnosis of pSS under consultation of the rheumatologists enrolled in the study will be included.
  Interventions: Other: PSC questionnaire

INTERVENTIONS:
Other: Interview — A one hour survey interview will be completed by the rheumatologists which will contain open and closed questions to probe physician perception and behaviors in relation to pSS management and treatment
  Groups: Physicians
Other: PSC questionnaire — All subjects for whom the physician completes a PRF will be required to complete a PSC questionnaire independently of their physician, immediately after consultation.
  Groups: Subjects with pSS
Other: PRFs — PRFs will be completed by the physicians for seven of their consulting pSS subjects.
  Groups: Physicians

SUMMARY:
Sjogren's Syndrome is a chronic autoimmune disease characterized by sicca (dryness) symptoms of the mouth and eyes. This autoimmune disease is less commonly studied and there are no licensed treatments to treat the underlying cause of disease and current management is based on clinical experience and/or small clinical studies. This study is based on DSP methodology, a multinational, cross-sectional, multi-sponsor survey of robust real-world data. DSP methodology collects quantitative market research data. The pSS DSP will survey a sample of approximately 230 to 325 rheumatologists and their prospectively consulting pSS subjects in France, Germany, Italy, Spain and the US. The data will be collected via physician interviews, physician workload questionnaires, detailed patient record forms (PRFs) to be completed by physicians, and a self-completion questionnaire by pSS subjects. The data collected using this method includes subjective and objective evidence, clinical information about individual patients, their disease and their treatment. This DSP will follow three key phases: preparatory phase, data collection phase and data processing/analysis phase.

ELIGIBILITY:
Inclusion Criteria:

Physician eligibility criteria:

* Primary physician specialty identified as Rheumatologist
* Physicians who currently treat 7 or more pSS subjects in a typical month
* Physicians who are actively involved in the management and treatment decisions of pSS subjects

Subject eligibility criteria:

* Subjects with a diagnosis of Sjogren's syndrome in the opinion of the rheumatologist in the absence of Systemic Lupus Erythematosus (SLE), Rheumatoid Arthritis (RA) or Systemic Sclerosis.
* For main sample (6 subjects per rheumatologist)
* Subjects with age >=18 years and with confirmed diagnosis of pSS and are currently, or have previously, exhibited disease activity in one or more of the categories: fever of non-infectious origin, lymphadenopathy/lymphoma, glandular swelling/enlarged parotid gland, arthralgia/synovitis, erythema/vasculitis/purpura, pulmonary involvement, renal involvement, myositis, peripheral nervous system involvement, central nervous system involvement, cytopenia of autoimmune origin (with neutropenia) and/or anemia and/or thrombocytopenia and/or lymphopenia, hypocomplementemia and/or hypergammaglobulinemia and/or cryoglobulinemia or hypogammaglobulinemia and/or Ever received immunosuppressant or biologic treatment.
* For oversample (1 subject per rheumatologist)
* Subjects with age >=18 years and with confirmed diagnosis of pSS that fit the following criteria: Has never exhibited disease activity in any of the categories above, Moderate or severe fatigue (in the opinion of the rheumatologist)

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 230-325 rheumatologists actively involved in management and treatment decisions of pSS subjects in France, Italy, Spain, Germany and the United States and their prospectively consulting subjects with a confirmed diagnosis of pSS will be included in the DSP.
Sampling Method: Non-Probability Sample
Enrollment: 2223 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Physician reported categorization of pSS subjects | Baseline
  The most common categorization of pSS subjects by rheumatologists will be described, alongside differences in humanistic and clinical burden of these categories.
Statistically derived clusters of pSS subjects | Baseline
  Subject clusters will be statistically derived from demographic, clinical and humanistic characteristics.

SECONDARY OUTCOMES:
Description of subject's journey | As reported
  Summary of subject's journeys from diagnosis to current management and treatment, including an overview of HCRU.
Drivers of physician and subject reported satisfaction | Baseline
  Data for drivers of physician and subjects reported satisfaction with disease activity control and symptomatic relief will be derived.
Level of concordance/discordance between physician and patient reported satisfaction | Baseline
  Data for discordance/concordance between physicians and subjects across key measures will be derived.
Differences in subjects journey, physician and subjects reported satisfaction amongst the clusters identified in the primary objective | As reported / Baseline
  Differences in subjects journey, physician and subjects reported satisfaction amongst the clusters identified in the primary objective will be described.
Physician experience of biologic therapy | Baseline
  Physicians' experience of biologic therapy, and attitudes towards biologic therapy for subjects with pSS will be described.
Physician perception of treatment targets | Baseline
  Physicians' perceptions of treatment targets in pSS will be described.
subjects attitude towards route of administration | Baseline
  Proportion of subjects willing to take medication by type of administration route (oral/tablet, subcutaneous injection, intravenously) will be described.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- Adelphi Real World Investigational Site, Cheshire, United Kingdom